CLINICAL TRIAL: NCT07007351
Title: Comparative, Prospective, Single-blinded, Randomized, Multi-Center Clinical Trial to Determine the Performance and Safety of a New Device Injectable Micro-filler Solution Based on Hyaluronic Acid M-HA®30 Architect on the Skin Quality of the Face, Neck and décolleté and Comparing to a Reference Product, Profhilo® on the Lower Part of the Face and Neck: HEBE 8 Study
Brief Title: Multicenter, Prospective Study to Determine the Performance and Safety of the New M-HA30 Architect Device on the Quality of the Skin: HEBE8 Study
Acronym: HEBE8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires FILLMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-A00173-40; CIV-22-09-040866 (Other: EUDAMED)
Record Dates: First submitted 2025-05-07; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Skin Aging
MeSH Terms: interventions — Injections, Intradermal

STUDY DESIGN:
Intervention Model Description: This is a split face study (the investigational product could be injected on the left or on the right); the comparator will be injected on the opposite side
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHA30 injected on the Left (Split face study) for Face and Neck (Décolleté is not comparative) (Experimental): In assessing the aesthetic performance and safety of devices, the inter-individual variability is very large. As a result, a methodology often used is split-face evaluation , the subject being its own control. Schematically, the area of application (right or left hemiface) is drawn randomly and evaluations are done separately. It is a single blind study: during the injections, the eyes of the subject will be obscured by 2 ocular pads. As the procedure of injection of Profhilo for the face does not include the forehead and crow's feet, comparison will be performed with this device only on the lower part of the face (only M-HA®30 Architect will be injected on the crow's feet and forehead for a non-comparative before-after evolution study).
  As wrinkles of the décolleté are present mainly in the center of the décolleté, it was decided not to make a comparative on this area (only M-HA®30 Architect will be injected).
  Interventions: Device: Intradermal injection
- MHA-30 injected on the Right (Split face study) for Face and Neck (Décolleté is not comparative) (Experimental): In assessing the aesthetic performance and safety of devices, the inter-individual variability is very large. As a result, a methodology often used is split-face evaluation , the subject being its own control. Schematically, the area of application (right or left hemiface) is drawn randomly and evaluations are done separately. It is a single blind study: during the injections, the eyes of the subject will be obscured by 2 ocular pads. As the procedure of injection of Profhilo for the face does not include the forehead and crow's feet, comparison will be performed with this device only on the lower part of the face (only M-HA®30 Architect will be injected on the crow's feet and forehead for a non-comparative before-after evolution study).
  As wrinkles of the décolleté are present mainly in the center of the décolleté, it was decided not to make a comparative on this area (only M-HA®30 Architect will be injected).
  Interventions: Device: Intradermal injection

INTERVENTIONS:
Device: Intradermal injection — The product is the first solution with free hyaluronic acid boosted with silicium the administration mode is same as any other intradermal multi-injection procedure

SUMMARY:
For skin rejuvenation the targeted population does not present a specific pathology. Aesthetic procedures are requested by the patient to improve appearance, look younger and feel better.

Non-crosslinked Hyaluronic acid (HA) is widely used by intradermal multiple injection as it is a glycosaminoglycan, which binds and retains water thus improving the wrinkles while the tone and elasticity of the skin.

Previous studies showed that an important administration of Si had benefic effects on bone development, skin ageing and fragile hair and nails.

The major issue of the Si intake is the rapid absorption and excretion, and consequently low effects on the skin. Moreover, with ageing, gastric pH become more acidic and decreases the conversion capacity of the Si.

All these data together led Laboratoires Fillmed to develop an HA product boosted by Si to inject into ther dermis in order to fill fine lines wrinkes and improve skin quality.

This study aims to demonstrate the efficacy of this new Hyaluronic Acid based filler versus a reference device, with an intradermal multi-injection technique, on reducing the superficial wrinkles measured by comparative evaluation between baseline and D30+10 of the evolution of wrinkles of the face / neck and décolleté by clinical scoring.

To this end, subjects in whom a correction of wrinkles of the face and/or décolleté and/or neck is sought, will be included. Subjects will receive 2 sessions of treatment on each side of the concerned area and the aesthetic correction will be appreciated at 10 ± 2 days (D30+10) following the last treatment session and the maintenance of the correction will be evaluated on D60, D120 and D180.

Main objective:

The main objective of this randomized study is to demonstrate objectively the effectiveness of the studied device, on the reduction of the universal wrinkles score, performed in presence of the subjects, between baseline and D30+10 (10 days after the last injection) on the cheeks, neck or décolleté and its non-inferiority by intraindividual comparison versus a reference device for the cheek and the neck.

Secondary objectives:

* For all groups and for the concerned zones:

  - to assess the efficacy of the devices between baseline and D180 (including D0, D30+10, D60, D120 and D180) and comparatively evaluate the efficacy for the cheeks and neck of the tested device compared to the reference device on:
* the Universal Wrinkles Score performed on the cheek's wrinkles, neck wrinkles or décolleté's wrinkles by the investigators, in presence of the subjects
* Zone-specific (cheek, neck or décolleté) clinical scores performed from photographical visual scales, Clinical score of radiance (for the face)
* the Universal Wrinkles Score performed at the end of the study in a blind manner by an expert on the cheek's wrinkles, neck wrinkles or décolleté's wrinkles from the standardized photographs

  - to assess the efficacy of the devices from D30 to D180 on the Global Aesthetic Improvement Scores performed by:
* the investigator (IGAIS) for 5 items
* the subjects (SGAIS) for 5 items

  * to assess the safety, efficacy and the opinion of the subjects by a questionnaire
  * to illustrate the efficacy of the devices by standardized photographs

Three Research Centerswere added to the study to have objective and instrumental data on the efficacy of the products on skin's:

* hydration by Corneometer®
* firmness and elasticity by CutoMeter®
* density by Ultrasound Imaging
* anatomical characteristics by in vivo Reflectance Confocal Microscopy
* anatomical characteristics by in vivo Optical Coherence Tomography
* the average volume of wrinkles (depth and surface) measured on the cheeks from image processing performed from 3D imaging

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects except for injections on the décolleté that will only concern women
2. From 19 to 84 years old
3. Who has signed a written informed consent;
4. With a Fitzpatrick phototype of I, II, III or IV
5. Having on both sides, one of the 3 following conditions:

   * For Face: a wrinkle score according to Lemperle scale of 2, 3 or 4 at the level of the cheeks
   * For Neck: a Grade 2, 3 or 4 on Bazin Neck Wrinkle Scale
   * For Decollte: a Grade 2 or 3 on Landau Décolleté Wrinkle Scale
6. Registered with Social Security (for France)
7. Accepting not to expose him/herself to the sun or ultraviolet (UV) during the entire duration of the study.
8. For female of childbearing potential accepting to take a pregnancy test (a pregnancy test will be performed before each injection) and a highly effective contraception* method during whole study.

Exclusion Criteria:

1. Subject involved in any other clinical study evaluating drugs or medical devices, including devices without an intended medical purpose, or subjects in exclusion periods of another clinical study.
2. Deprived of freedom by an administrative or legal decision.
3. Unable to follow protocol requirements.
4. Who has received compensation of 4500 € during the 12 previous months for his/her participation in clinical trials (including participation in this study / for France).
5. Having benefit from injection/facial implantation of any non-absorbable filling agent at any time of his/her life.
6. Having already had laser sessions for skin rejuvenation or a laser facelift in the previous year or a facelift by surgery in the 2 years prior to the study.
7. With a history of absorbable fillers injections (such as hyaluronic acid) in the last year or botulinum toxin in the last 6 months or the injectable implants (semi-permanent fillers) in the last two years.
8. With a skin support device (wire mesh, gold wire, liquid silicone or other particulate material, absorbable or non-absorbable threads) at the study zones.
9. Having done a moderate to deep peeling or non-invasive rejuvenation techniques such as radiofrequency, ultrasound and lasers in the last 6 months.
10. With a history of multiple severe allergies or anaphylactic shock.
11. With a known hypersensitivity to hyaluronic acid, or other components of M-HA®30 Architect and Profhilo®.
12. With a known hypersensitivity to the disinfection products such as chlorhexidine and betadine.
13. With a known hypersensitivity to lidocaine or to local amide-type anesthetics.
14. Prone to developing inflammatory skin conditions or hypertrophic scarring according to investigator judgement.
15. With a history of streptococcal diseases (angina recurrent, rheumatic fever).
16. Under concomitant treatment (or not stopped for at least 3 months) by oral or injectable corticosteroid (inhaled corticosteroids are allowed as well as a topical corticotherapy not involving the study zones).
17. Under concomitant treatment (or not stopped for at least 1 year) by immunosuppressive or chemotherapy treatments.
18. With a history of less than one year of radiation therapy in the investigated areas.
19. With an associated antecedent or pathology of autoimmune or connective tissue disease.
20. Presenting a skin pathology, an acute inflammatory reaction or a bacterial or viral infection on the study zones or within the 6 weeks after the end of such an episode.
21. With heart disease and/or undergoing treatment for heart disease (beta-blockers)
22. With congenital glucose-6-phosphate dehydrogenase deficiency or idiopathic methemoglobinemia
23. With hepatocellular insufficiency and/or undergoing treatment for liver disease
24. With porphyria
25. Having taken aspirin or anticoagulants, at regular doses, in the last 15 days preceding the act.
26. That has been exposed to sun or UV in the last 15 days.
27. With a dermatological condition or inflammation at the treatment zone or near to this area (according to the investigator's judgment).
28. Pregnant or lactating woman (Before every injection, a urinary pregnancy test will be performed).
29. Having epilepsy uncontrolled by treatment.
30. Presenting a general pathology, skin pathology, dermatosis, systemic, chronic or acute disease and/or topical or general treatment that in the opinion of the investigator may interfere with the treatment or compromise the participation of the subject in the study.
31. With a COVID vaccination plan of any dose with any kind of vaccine at 3 weeks before or 3 weeks after each injection session.
32. With a history of COVID infection in the last 4 weeks and still have a positive test and/or the raised inflammatory markers such as ferritin, CRP, IL-8, D-Dimer, etc. (blood results will only be requested for volunteers with a severe form of the disease, i.e. one that required medical intervention or hospitalization).

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2023-03-19 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Universal wrinkles score | Between Day 0 and Day 40
  Universal Wrinkles Score (UWS) inspired from the Modified Fitzpatrick Wrinkles Scale. It is a 7 grades score.
  Score definition 0 No wrinkle
  1. Very shallow wrinkle
  2. Fine wrinkle
  3. Fine to moderate wrinkles
  4. Moderate wrinkle
  5. Deep wrinkle
  6. Very deep wrinkle

CONTACTS AND LOCATIONS:
Locations (1):
- Fillmed Laboratoires, Paris, France